CLINICAL TRIAL: NCT00168857
Title: A Prospective, Randomised, Double-blind, Double-dummy, Forced-titration, Multicentre, Parallel Group, One Year Treatment Trial to Compare MICARDIS® (Telmisartan) 80 mg Versus COZAAR® (Losartan) 100 mg, in Hypertensive Type 2 Diabetic Patients With Overt Nephropathy (AMADEO Study)
Brief Title: A Prospective, Randomised, Double-blind, Double-dummy, Forced-titration, Multicentre, Parallel Group, One Year Treatment Trial to Compare Telmisartan (MICARDIS) 80 mg Versus Losartan (COZAAR) 100 mg, in Hypertensive Type 2 Diabetic Patients With Overt Nephropathy (AMADEO Study)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.397
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Diabetic Nephropathies
MeSH Terms: conditions — Hypertension; Diabetic Nephropathies | interventions — Telmisartan; Losartan

INTERVENTIONS:
Drug: telmisartan
Drug: losartan

SUMMARY:
A number of blood pressure lowering drugs in the class known as angiotensin receptor blockers (ARB) have been shown to slow the decline in kidney function of patients with type 2 diabetes, high blood pressure, and kidney disease. Losartan (COZAAR), is one such drug. The purpose of this research study is to determine if after one year of treatment telmisartan (MICARDIS, GLIOSARTAN, KINZAL, KINZALMONO, PREDXAL, PRITOR, SAMERTAN, TELMISARTAN) 80 mg, another blood pressure lowering drug from the ARB class, is as effective as losartan (COZAAR) 100 mg in reducing the level of urinary protein (indicative of improved kidney function).

ELIGIBILITY:
Inclusion criteria:

* Ability to provide written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age 21-80 years
* Clinical history of type 2 diabetes mellitus, as defined by either:

  * Hyperglycaemia not requiring insulin (diet, oral hypoglycaemic agents and metformin if patients serum creatinine levels were within normal limits.)
  * Hyperglycaemia requiring insulin with: no history of diabetic ketoacidosis AND with either the period between diagnosis and insulin usage >1 year or elevated fasting or stimulated C-peptide level
* Glycosylated haemoglobin A1 (HbA1c) ≤10%
* Diabetic nephropathy, as defined by:

  * serum creatinine at Screening (Visit 1) ≤265 μmol/L (3.0 mg/dL) in women and ≤283 μmol/L (3.2 mg/dL) in men
  * urinary protein/creatinine ratio ≥700 mg/g (measured in spot urine) during the run-in phase (Visit 2 or Visit 5 retest)
* Hypertension at screening, as defined by either:

  * Mean systolic blood pressure (SBP) >130 mmHg and/or mean diastolic blood pressure (DBP) >80 mmHg in untreated patients
  * Patients currently receiving antihypertensive medication (i.e. medications specifically prescribed to treat hypertension)
* Ability to stop current antihypertensive therapy with Angiotensin Converting Enzyme Inhibitor (ACE-Is), Angiotensin Receptor Blockers (ARBs) and direct vasodilators, and to stop chronic immunosuppressive therapy and current therapy with metformin without risk to the patient (Investigator's discretion).
* All female patients had to have negative results from the urine pregnancy test (UPT) at Visits 1 and 6 in order to be able to continue in the study.

Exclusion criteria:

* Pre-menopausal women (last menstruation ≤1 year prior to signing informed consent) who:

  * were not surgically sterile or
  * were nursing or pregnant or
  * were of child-bearing potential and were not practicing acceptable methods of birth control, or did not plan to continue practicing an acceptable method throughout the study (Note: Acceptable methods of birth control included transdermal patch, intra-uterine device, oral, implantable or injectable contraceptives) AND did not agree to periodic urine pregnancy testing (UPT) during participation in the study. No exceptions were made.
* Type 1 diabetes mellitus
* Increase of serum creatinine >35% between Visit 1 (Screening) and Visit 5. If creatinine was increased >35% at Visit 5, the measurement was to be repeated within five calendar days and if the increase was confirmed, the patient had to be excluded from the trial for safety reasons.
* Non-diabetic renal disease
* Congestive heart failure (New York Heart Association functional class III or IV)
* Unstable angina, myocardial infarction, coronary artery bypass graft surgery, or percutaneous coronary intervention within the last three months prior to signing the informed consent form
* Stroke or transient ischaemic attack within the last six months prior to signing the informed consent form
* Hypertrophic obstructive cardiomyopathy, hemodynamically relevant stenosis of the aortic or mitral valve
* Further exclusion criteria apply

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 860 (Actual)
Dates: Start 2003-07-09 (Actual); Primary Completion 2006-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline after one year of treatment in proteinuria (ratio of protein to creatinine as measure in spot urine sample). | Up to 1 year

SECONDARY OUTCOMES:
Change from baseline after one year of treatment in the following: glomerular filtration rate; serum creatinine; macroalbuminuria; sodium excretion; high sensitive C-reactive protein; serum aldosterone; and other renal and cardiovascular measures. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (109):
- United States (47):
  - Boehringer Ingelheim Investigational Site, Montgomery, Alabama
  - Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - Boehringer Ingelheim Investigational Site, Lancaster, California
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - VA of Greater Los Angeles, Los Angeles, California
  - UCI Medical Center, Orange, California
  - VA San Diego Healthcare System, San Diego, California
  - Boehringer Ingelheim Investigational Site, Santa Ana, California
  - UCLA Medical Center, Sylmar, California
  - Torrance Clinical Research, Torrance, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - George Washington University, Washington D.C., District of Columbia
  - Boehringer Ingelheim Investigational Site, Hollywood, Florida
  - Boehringer Ingelheim Investigational Site, Largo, Florida
  - Boehringer Ingelheim Investigational Site, Ocala, Florida
  - Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - Boehringer Ingelheim Investigational Site, Tampa, Florida
  - Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush Presbyterian - St. Lukes Medical Center, Chicago, Illinois
  - Boehringer Ingelheim Investigational Site, Des Moines, Iowa
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - Boehringer Ingelheim Investigational Site, Towson, Maryland
  - Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - Boehringer Ingelheim Investigational Site, Eatontown, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Boehringer Ingelheim Investigational Site, Flushing, New York
  - Winthrop University Hospital, Mineola, New York
  - Harlem Hospital, New York, New York
  - Northport VAMC - Medical Service (111), Northport, New York
  - Wake Nephrology Associates, PA, Raleigh, North Carolina
  - The Cleveland Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - University of Texas Health and Science Center at San Antonio, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - University of Virginia Health Science Center, Charlottesville, Virginia
  - Boehringer Ingelheim Investigational Site, Gig Harbor, Washington
  - Boehringer Ingelheim Investigational Site, Seattle, Washington
  - Clement J. Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
- Argentina (8):
  - Boehringer Ingelheim Investigational Site, Buenos Aires
  - Clinica Coronel Suarez, Coronel Suárez
  - Boehringer Ingelheim Investigational Site, Córdoba
  - Boehringer Ingelheim Investigational Site, Paraná
  - Boehringer Ingelheim Investigational Site, Provincia de Buenos Aires
  - Boehringer Ingelheim Investigational Site, Rosario, Santa Fé
  - Hospital San Bernardo, Salta
  - Boehringer Ingelheim Investigational Site, Santa Fe
- Australia (4):
  - Boehringer Ingelheim Investigational Site, Kippa-Ring, Queensland
  - Lyell McEwin Hospital Department of medicine, Elizabeth, South Australia
  - Geelong Clinical Research Centre, Geelong, Victoria
  - Boehringer Ingelheim Investigational Site, Melbourne, Victoria
- Brazil (4):
  - Universidade Federal do Pará, Belém
  - Boehringer Ingelheim Investigational Site, Botucatu
  - Faculdade de Medicina Universidade Federal de Juiz de Fora, Juiz de Fora ¿ MG
  - Boehringer Ingelheim Investigational Site, Vila Clementino, São Paulo
- Canada (22):
  - Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - Boehringer Ingelheim Investigational Site, Red Deer, Alberta
  - BC Endocrine Research Foundation, Vancouver, British Columbia
  - Endocrine Research Society, Vancouver, British Columbia
  - University of Manitoba, Diabetes Research Group, Winnipeg, Manitoba
  - Division of Respirology, Halifax, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Kitchener, Ontario
  - Boehringer Ingelheim Investigational Site, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, Oakville, Ontario
  - The Ottawa Hospital - Riverside Campus, Ottawa, Ontario
  - LIfestyle Metabolism Centre - Thornhill, Thornhill, Ontario
  - Boehringer Ingelheim Investigational Site, Timmins, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook & Woman's College Health Science Centre, Toronto, Ontario
  - Humber River Regional Hospital, Dialysis Unit, Weston, Ontario
  - Boehringer Ingelheim Investigational Site, Laval, Quebec
  - CHUM - Hote-Dieu, Montreal, Quebec
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - CHUS - Hopital Fleurimont, Sherbrooke, Quebec
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Mexico (7):
  - Fracc. Magallanes, Acapulco Guerrero
  - Boehringer Ingelheim Investigational Site, Col. Sección XVI, Deleg. Tlalpan
  - Cardiology, Guadalajara
  - Hospital Civil Nuevo de Guadalajara, Guadalajara
  - Boehringer Ingelheim Investigational Site, Guadalajara, Jalisco
  - Dep of Neurology, Metepec
  - Cardiologia, México, D.F.
- New Zealand (2):
  - Boehringer Ingelheim Investigational Site, Auckland
  - 1st Floor Hagely Hostel, Christchurch
- South Korea (3):
  - Dongsan Medical Center, Daegu
  - National Health Insurance Corporation, Ilsan Hospital, Gyunggido
  - Yongdong Severance Hospital, Seoul
- Taiwan (6):
  - Buddhist Tzu Chi General Hospital, Chiayi City
  - Buddhist Tzu Chi General Hospital, Hualien City
  - Chi Mei Medical Center, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (6):
  - Bumrungrad Hospital, Bangkok
  - Pramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Division of Hypertension, Bangkok
  - Thummasart University Hospital, Bangkok
  - Maharaj Nakom Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Bakris G, Burgess E, Weir M, Davidai G, Koval S; AMADEO Study Investigators. Telmisartan is more effective than losartan in reducing proteinuria in patients with diabetic nephropathy. Kidney Int. 2008 Aug;74(3):364-9. doi: 10.1038/ki.2008.204. Epub 2008 May 21. PMID 18496508